CLINICAL TRIAL: NCT02337647
Title: Evaluation of the Distortion Correction Data Collection (DCDC) App Software to Repair Visual Distortions for Low Vision Age-related Macular Degeneration, and the Correlation of the Distortions With Clinical Examination
Brief Title: Evaluation of the Distortion Correction Data Collection (DCDC) App Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0625-14-FB
Record Dates: First submitted 2014-12-17; First posted 2015-01-13 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCDC app (Other): Subjects will evaluate the DCDC app
  Interventions: Other: DCDC App

INTERVENTIONS:
Other: DCDC App — The DCDC app is an experimental software that allows users to map their visual distortions on a tablet computer.

SUMMARY:
The purpose of the research study is to evaluate how well the Distortion Correction Data Collection (DCDC) App works. The DCDC App is an experimental software application that is being developed at the University of Nebraska Omaha. The DCDC app will map and draw the visual distortions of patients with Age-related Macular degeneration.

DETAILED DESCRIPTION:
This research study is a phase 1 clinical trial to evaluate the efficacy of the Distortion Correction Data Collection (DCDC) App on a computer tablet system. There are two objectives in this study. The primary objective is to evaluate the functionality of the visual distortion app on the tablet computer. Patients will draw their distortions on the tablet screen, and the app will record and correct the distortions.The second objective is to create a distortion data repository (DDR) that contains retinal maps, data pertaining to the anatomical and functional aspects of patients retinas and the distortions. This DDR will be used to correlate retinal health to distortions.The correlation will be key in improving the correction software of the app. Long term, the app will be used to create a diagnostic tool and improve image processing in retinal prosthesis systems.

Participating subjects must be at least 55 years of age or older with age-related macular degeneration (AMD). After consent, a chart review will be performed. At the baseline visit, subjects will have an electroretinogram (ERG). At the single study visit, to be scheduled within 2 weeks of the baseline visit, subjects will use the DCDC app on a tablet computer to trace their visual distortions on an Amsler grid. Up to 5 subjects who meet the inclusion/exclusion criteria will be enrolled. The duration of the study is a 2 hour baseline visit and a 1 hour study visit, all within 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or greater
* Diagnosed with age-related macular degeneration (AMD).
* Best corrected visual acuity (BCVA) of (20/40 to 20/200 Snellen equivalent).
* Visual distortion is present in at least one eye, as determined by Amsler grid evaluation.
* Have had the following imaging tests completed within the past three months as part of standard of care: optical coherence tomography (OCT), scanning laser ophthalmoscopy (SLO), and Fluorescein angiography (FA).
* Capable of understanding the requirements of the study, willing to follow study instructions, able to provide written informed consent to participate, and willing to comply with all study requirements.
* Women who are post-menopausal or not otherwise of child-bearing potential -

Exclusion Criteria:

* Visual field loss from diseases other than AMD.
* Visual distortions from the following conditions other than AMD: epiretinal membrane, diabetic macular edema, central retinal vein occlusion (CRVO) with edema, and cystoid macular edema.
* A medical condition, serious concurrent illness, or extenuating circumstance that would significantly decrease ability to follow study instructions.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Functionality of the Distortion Correction Data Collection App (DCDC), as measured by successful usage of the app by subjects. | 3 months
  Subjects will use the app to trace visual distortions. The app will correct these distortions, subjects will give feedback on these corrections. Test will be repeated two times.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gulati, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Truhlsen Eye Institute, Omaha, Nebraska, United States